CLINICAL TRIAL: NCT06541912
Title: Comparative Evaluation of Implant Stability, Soft and Hard Tissue Healing Around UV Activated Versus Conventional Implants - A Randomized Clinical Trial.
Brief Title: Comparative Evaluation of Implant Stability, Soft & Hard Tissue Healing Around UV Activated vs Conventional Implants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 02_D012_00048
Record Dates: First submitted 2024-07-19; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: UV Dental Implant
Keywords: Dental Implants
MeSH Terms: interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional dental implant group (Active Comparator): conventional dental implant placement will act as control group.
  Interventions: Procedure: conventional implant
- UV dental implant group (Experimental): UV activated implant placement will act as test group which has better osseointegration properties.
  Interventions: Procedure: UV implant

INTERVENTIONS:
Procedure: conventional implant — A full thickness mucoperiosteal flap was elevated under local anesthesia, osteotomy sites were prepared according to manufacturer's instructions and parallel pin was used to confirm position and angulation of osteotomy site. Conventional implant placement was done on one side.
  Resonance frequency analysis instrument was used to measure Implant Stability Quotient (ISQ) and check the primary stability of the implant. The surgical wound closure was done with mattress and single interrupted sutures, using 4-0 vicryl sutures.
  Arms: conventional dental implant group
Procedure: UV implant — A full thickness mucoperiosteal flap was elevated under local anesthesia and osteotomy sites were prepared according to manufacturer's instructions. Parallel pin was used to confirm position and angulation of osteotomy site. UV implant was activated using UV Activator2 and placed in another site.
  Resonance frequency analysis instrument was used to measure Implant Stability Quotient (ISQ) and primary stability of the implant was measured. The surgical wound closure was done with mattress and single interrupted sutures, using 4-0 vicryl sutures.
  Arms: UV dental implant group

SUMMARY:
Research is to compare and evaluate the primary and secondary implant stability, healing of the soft tissue around UV activated implants and conventional implants.

DETAILED DESCRIPTION:
Research is to compare and evaluate the primary and secondary implant stability, healing of the soft tissue around UV activated implants and conventional implants. The objectives are to access the primary and secondary implant stability using Resonance frequency analysis, marginal bone level using RVG with grid, healing of the soft tissue. The control group will be treated with conventional implant and test group will be treated with UV implants. The total number of participants are 12 and 24 sites (control - 12 sites, test - 12 sites) with 3 months follow up.

ELIGIBILITY:
Inclusion Criteria:

* At east above 18 years of age
* Patients who needs replacement for at least 2 missing teeth in the posterior region of mandible
* Adequate bone volume to accommodate planned dental implants
* Patients who will comply with oral health care instructions and necessary visits

Exclusion Criteria:

* General contraindications to dental implant treatment ( uncontrolled diabetes, severe cardiovascular or infectious disease)
* Intravenous and oral bisphosphonate therapy
* Unwillingness to return for the follow up examinations
* Smokers
* Patients who are psychologically unable to participate
* Poor oral hygiene

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-03-25 (Estimated)

PRIMARY OUTCOMES:
Implant stability using Resonance Frequency Analysis | "Immediately after Post-operative", "1 month", "3 months"
  to measure primary and secondary stability

SECONDARY OUTCOMES:
Marginal bone loss using RVG with grid | "Immediately after Post-operative", 3 months
  to measure marginal bone level
Soft tissue healing | 1 week, 1 month, 3 months.
  soft tissue healing to be assessed using Landry Turnbull and Howley Healing Index. Soft tissue healing will be scored from 1 to 5, where score 1 is very poor and 5 is excellent.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Prabhuji MLV, Bengaluru, Karnataka, India